CLINICAL TRIAL: NCT03481309
Title: Modulation of Motor Cortex Excitability by Transcranial Magnetic Stimulation and Transcranial Direct Current Stimulation
Brief Title: Modulation of Motor Cortex Excitability by TMS and tDCS (MAGS1)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 17-0149; R01MH101547 (NIH)
Record Dates: First submitted 2018-03-09; First posted 2018-03-29 (Actual); Results first posted 2019-10-23 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Motor Activity; Motor Neuroplasticity
Keywords: transcranial magnetic stimulation (TMS); transcranial direct current stimulation (tDCS); electroencephalography (EEG)
MeSH Terms: conditions — Motor Activity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Each participant will be assigned to 2 active and sham conditions on a different day.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind and cross-over study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- anodal tDCS (Active Comparator): Two electrodes will be applied to the scalp (one on the left motor cortex, one on the right supraorbital cortex). This anodal tDCS on the left motor cortex will be stimulated with 2mA for 10 minutes.
  Interventions: Device: anodal tDCS
- cathodal tDCS (Active Comparator): Two electrodes will be applied to the scalp (one on the left motor cortex, one on the right supraorbital cortex). This cathodal tDCS on the left motor cortex will be stimulated with -2mA for 10 minutes.
  Interventions: Device: cathodal tDCS
- sham tDCS (Sham Comparator): Two electrodes will be applied to the scalp (one on the left motor cortex, one on the right supraorbital cortex). Sham stimulation with 2mA for 40 seconds will be applied.
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: anodal tDCS — The participant will receive anodal tDCS with 2 mA for 10 minutes on the left motor cortex.
  Arms: anodal tDCS
Device: cathodal tDCS — The participant will receive cathodal tDCS with -2 mA for 10 minutes on the left motor cortex.
  Arms: cathodal tDCS
Device: sham tDCS — The participant will receive sham tDCS with 2 mA for 40 seconds on the left motor cortex which mimics the skin sensations as active tDCS interventions.
  Arms: sham tDCS

SUMMARY:
Investigating modulation of motor cortex excitability by transcranial magnetic stimulation and transcranial direct current stimulation.

DETAILED DESCRIPTION:
Purpose of this pilot study is to modulate the motor cortex excitability by transcranial magnetic stimulation and transcranial direct current stimulation. Electromyography will be recorded on right abductor digiti minimi muscle to find the motor threshold and measure motor evoked potentials for each healthy participant. In addition, electroencephalography (EEG) data will be collected on the scalp with a high-density EEG net. Eighteen healthy participants will be in this study. Each participant will be seated in a reclining chair and applied non-invasive magnetic and electrical stimulations on the scalp. At baseline, the participant's resting motor threshold (RMT) will be estimated by adjusting the intensity of TMS applied on the left motor cortex to achieve motor-evoked potentials of about 50 uV with 10 TMS pulses at a rate of 0.25 Hz. Then a 3-condition, 3-session, 6-sequence randomized crossover experiment will be used to characterize and compare three versions of tDCS stimulation: anode, cathode, sham. Before and after a 10-min tDCS condition is applied, TMS pulses at 120% of RMT intensity will be applied for 10 minutes and TMS-evoked potential and motor-evoked potential amplitudes will be measured. Each session has at least 1-day gap to remove outlasting effects. We will also be collecting structural magnetic resonance imaging (sMRI) to target primary motor cortex precisely.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Between the ages of 18 and 35
* Right-handed
* Capacity to understand all relevant risks and potential benefits of the study (informed consent)
* Willing to comply with all study procedures and be available for the duration of the study
* Speak and understand English

Exclusion Criteria:

* Prior concussion
* Diagnosis of eating disorder (current or within the past 6 months)
* Diagnosis of obsessive compulsive disorder (lifetime)
* Attention-deficit/hyperactivity disorder (currently under treatment)
* Neurological disorders and conditions, including, but not limited to:

  * History of epilepsy
  * Seizures (except childhood febrile seizures and electroconvulsive therapy-induced seizures)
  * Dementia
  * History of stroke
  * Parkinson's disease
  * Multiple sclerosis
  * Cerebral aneurysm
  * Brain tumors
* Medical or neurological illness or treatment for a medical disorder that could interfere with study participation (e.g., unstable cardiac disease, HIV/AIDS, malignancy, liver or renal impairment)
* Prior brain surgery
* Any brain devices/implants, including cochlear implants and aneurysm clips
* Traumatic brain injury
* Anything that, in the opinion of the investigator, would place the participant at increased risk or preclude the participant's full compliance with or completion of the study

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, Principal Investigator — University of North Carolina at Chapel Hill - Department of Psychiatry
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Anode -> Cathode -> Sham: During 3 study visits, participants will receive anodal tDCS first, then cathodal tDCS, then sham tDCS. For all three tDCS conditions, two electrodes will be applied to the scalp (one on the left motor cortex, one on the right supraorbital cortex) for 10 minutes.
- Anode -> Sham -> Cathode: During 3 study visits, participants will receive anodal tDCS first, then sham tDCS, then cathodal tDCS. For all three tDCS conditions, two electrodes will be applied to the scalp (one on the left motor cortex, one on the right supraorbital cortex) for 10 minutes.
- Cathode -> Anode -> Sham: During 3 study visits, participants will receive cathodal tDCS first, then anodal tDCS, then sham tDCS. For all three tDCS conditions, two electrodes will be applied to the scalp (one on the left motor cortex, one on the right supraorbital cortex) for 10 minutes.
- Cathode -> Sham -> Anode: During 3 study visits, participants will receive cathodal tDCS first, then sham tDCS, then anodal tDCS. For all three tDCS conditions, two electrodes will be applied to the scalp (one on the left motor cortex, one on the right supraorbital cortex) for 10 minutes.
- Sham -> Anode -> Cathode: During 3 study visits, participants will receive sham tDCS first, then anodal tDCS, then cathodal tDCS. For all three tDCS conditions, two electrodes will be applied to the scalp (one on the left motor cortex, one on the right supraorbital cortex) for 10 minutes.
- Sham -> Cathode -> Anode: During 3 study visits, participants will receive sham tDCS first, then cathodal tDCS, then anodal tDCS. For all three tDCS conditions, two electrodes will be applied to the scalp (one on the left motor cortex, one on the right supraorbital cortex) for 10 minutes.
Period: First Intervention (1 Day)
Arm/Group | Anode -> Cathode -> Sham | Anode -> Sham -> Cathode | Cathode -> Anode -> Sham | Cathode -> Sham -> Anode | Sham -> Anode -> Cathode | Sham -> Cathode -> Anode
Started | 4 | 3 | 3 | 3 | 3 | 3
Completed | 4 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (at Least 3 Days)
Arm/Group | Anode -> Cathode -> Sham | Anode -> Sham -> Cathode | Cathode -> Anode -> Sham | Cathode -> Sham -> Anode | Sham -> Anode -> Cathode | Sham -> Cathode -> Anode
Started | 4 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Anode -> Cathode -> Sham | Anode -> Sham -> Cathode | Cathode -> Anode -> Sham | Cathode -> Sham -> Anode | Sham -> Anode -> Cathode | Sham -> Cathode -> Anode
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (at Least 3 Days)
Arm/Group | Anode -> Cathode -> Sham | Anode -> Sham -> Cathode | Cathode -> Anode -> Sham | Cathode -> Sham -> Anode | Sham -> Anode -> Cathode | Sham -> Cathode -> Anode
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (1 Day)
Arm/Group | Anode -> Cathode -> Sham | Anode -> Sham -> Cathode | Cathode -> Anode -> Sham | Cathode -> Sham -> Anode | Sham -> Anode -> Cathode | Sham -> Cathode -> Anode
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One participant signed the consent form and provided baseline characteristics but research data collection for this participant was not performed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Anode -> Cathode -> Sham | Anode -> Sham -> Cathode | Cathode -> Anode -> Sham | Cathode -> Sham -> Anode | Sham -> Anode -> Cathode | Sham -> Cathode -> Anode | Total
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 3 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 3 | 3 | 3 | 3 | 19
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.75 (6.68) | 25.33 (6.94) | 22.33 (1.24) | 20.66 (0.47) | 22 (4.24) | 25.33 (6.12) | 24.31 (5.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 4 | 3 | 3 | 3 | 3 | 3 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 2 | 1 | 0 | 4
  White | 2 | 2 | 1 | 1 | 1 | 1 | 8
  More than one race | 1 | 1 | 1 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 3 | 3 | 3 | 3 | 19

OUTCOME MEASURES:

1. Primary Outcome: Changes in Motor-evoked Potentials Ratios
Description: The investigators will record motor-evoked potentials and calculate changes in between before and after 2mA tDCS stimulation for 10 minutes.
Time Frame: right before and after 2mA tDCS stimulation for 10 minutes at each session
Population: One participant signed the consent form but data for this participant was not recorded.
Measure: Mean (Standard Error); unit: Ratio (unit: uV)
Arm/Group | Anodal tDCS | Cathodal tDCS | Sham tDCS
Number analyzed (Participants) | 18 | 18 | 18
Ratio (unit: uV) | 1.32 (0.09) | 0.73 (0.07) | 1.03 (0.05)

2. Primary Outcome: Changes in TMS-evoked Potentials Ratios
Description: The investigators will record TMS-evoked potentials using EEG and calculate changes in between before and after 2mA tDCS stimulation for 10 minutes.
Time Frame: right before and after 2mA tDCS stimulation for 10 minutes at each session
Population: One participant signed the consent form but data for this participant was not recorded.
Measure: Mean (Standard Deviation); unit: Ratio (unit: uV)
Arm/Group | Anodal tDCS | Cathodal tDCS | Sham tDCS
Number analyzed (Participants) | 18 | 18 | 18
Ratio (unit: uV) | 1.5 (0.5) | 0.8 (0.4) | 1.1 (0.4)

3. Secondary Outcome: Changes in Resting-state EEG Dynamics Ratios
Description: The investigators will record participants' resting state for 4 minutes using EEG (2 minutes for eyes-closed and 2 minutes for eyes-open)
Time Frame: 4 minutes recordings before and after each 2mA tDCS stimulation for 10 minutes at each session
Population: One participant signed the consent form but data for this participant was not recorded.
Measure: Mean (Standard Deviation); unit: Ratio (unit: uV)
Arm/Group | Anodal tDCS | Cathodal tDCS | Sham tDCS
Number analyzed (Participants) | 18 | 18 | 18
Ratio (unit: uV) | 1.2 (0.7) | 0.8 (0.3) | 1.1 (0.5)

ADVERSE EVENTS:
Time Frame: After the study session on each day, an intervention was given, approximately 2 hours
Description: A side effects questionnaire
Arm/Group | Anodal tDCS | Cathodal tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/09/NCT03481309/Prot_SAP_000.pdf